CLINICAL TRIAL: NCT03860844
Title: Open-label, Single-arm Trial to Evaluate Antitumor Activity, Safety, and Pharmacokinetics of Isatuximab Used in Combination With Chemotherapy in Pediatric Patients From 28 Days to Less Than 18 Years of Age With Relapsed/Refractory B or T Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia in First or Second Relapse
Brief Title: Isatuximab in Combination With Chemotherapy in Pediatric Patients With Relapsed/Refractory Acute Lymphoblastic Leukemia or Acute Myeloid Leukemia
Acronym: ISAKIDS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was prematurely stopped due to sponsor decision (stage 2 efficacy criteria not met); not due to safety concerns.
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACT15378; PIP - 2018-002697-45; U1111-1202-1096 (Other: UTN); 2018-002697-45 (EudraCT Number)
Record Dates: First submitted 2019-02-21; First posted 2019-03-04 (Actual); Results first posted 2023-11-15 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
Keywords: Anti-CD38 monoclonal antibody
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — isatuximab; Dexamethasone; fludarabine; Cytarabine; Daunorubicin; Idarubicin; Filgrastim; Mitoxantrone; Doxorubicin; Vincristine; pegaspargase; Asparaginase; Cyclophosphamide; Etoposide; Methotrexate; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acute Myeloid Leukemia (AML) and Acute Lymphoblastic Leukemia (Experimental): This arm includes participants from 3 cohorts: AML, T-ALL and B-ALL.; AML: Weekly dosing of isatuximab with induction chemotherapy. The therapy may be repeated one more cycle; ALL: (Includes T-ALL and B-ALL) Weekly dosing of isatuximab with induction chemotherapy, then biweekly dosing of isatuximab with consolidation chemotherapy.
  Interventions: Drug: Isatuximab; Drug: Dexamethasone or equivalent; Drug: Fludarabine; Drug: Cytarabine; Drug: Liposomal daunorubicin; Drug: Daunorubicin (nonliposomal); Drug: Idarubicin; Drug: Filgrastim or equivalent; Drug: Mitoxantrone; Drug: Doxorubicin; Drug: Vincristine; Drug: Pegaspargase (PEG) Asparaginase; Drug: Cyclophosphamide; Drug: Etoposide; Drug: Methotrexate; Drug: L - Asparginase; Drug: Hydroxyurea; Drug: L - Asparaginase (Erwinase)

INTERVENTIONS:
Drug: Isatuximab — Pharmaceutical form: Concentrate for solution for intravenous infusion Route of administration: Intravenous
  Other Names: SAR650984; Sarclisa
Drug: Dexamethasone or equivalent — Pharmaceutical form: Solution for injection or tablet Route of administration: Intravenous or oral
Drug: Fludarabine — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Cytarabine — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Liposomal daunorubicin — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Daunorubicin (nonliposomal) — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
Drug: Idarubicin — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Filgrastim or equivalent — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Mitoxantrone — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Doxorubicin — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Vincristine — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Pegaspargase (PEG) Asparaginase — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
Drug: Cyclophosphamide — Pharmaceutical form: Solution for injection Route of administration: Intravenous
Drug: Etoposide — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
Drug: Methotrexate — Pharmaceutical form: Solution for injection Route of administration: Intravenous infusion
Drug: L - Asparginase — Pharmaceutical form: Solution for injection Route of administration: Intramuscular
Drug: Hydroxyurea — Pharmaceutical form: Solution for injection Route of administration: PO
Drug: L - Asparaginase (Erwinase) — Pharmaceutical form: Solution for injection Route of administration: Intramuscular

SUMMARY:
Primary Objective:

Evaluate the anti-leukemic activity of isatuximab in combination with standard chemotherapies in pediatric participants of ages 28 days to less than 18 years with Relapsed/Refractory Acute Lymphoblastic Leukemia (ALL) or Acute Myeloid Leukemia (AML)

Secondary Objectives:

* Safety and tolerability assessments
* Assessment of infusion reactions (IRs)
* Pharmacokinetics (PK) of isatuximab
* Minimal residual disease
* Overall response rate
* Overall survival
* Event free survival
* Duration of response
* Relationship between clinical effects and CD38 receptor density and occupancy

DETAILED DESCRIPTION:
The study included:

* a screening period of up to (up to 3 weeks prior to the first study treatment administration);
* a study treatment period [Day 1 to Day 57 for Acute Lymphoblastic Leukemia (ALL); Day 1 to Day 22 for Acute Myeloid Leukemia (AML)];
* the period of aplasia followed by a recovery period;
* an end of treatment (EOT) visit [within 30 days after hematological recovery;
* a follow-up period (until final analysis cut off date).

ELIGIBILITY:
Inclusion criteria:

* Participant 28 days to less than 18 years of age, at the time of signing the informed consent.
* Participants must have had a confirmed diagnosis of relapsed Acute Lymphoblastic Leukemia (ALL) of T- or B-cell origin including T-lymphoblastic lymphoma (LBL), or relapsed Acute Myeloblastic Leukemia (AML) including participants with history of myelodysplasia.
* Participants must have been previously treated for their disease and have relapsed or are refractory to most recent treatment. Participants in first or second relapse were eligible regardless of the remission duration.
* Participants who had no more than 1 prior salvage therapy.
* White Blood Cell (WBC) counts below 20 x10^9/L on Day 1 before isatuximab administration

Exclusion criteria:

* Any serious active disease or co-morbid condition which, in the opinion of the Investigator, may interfere with the safety of the study treatment or the compliance with the study protocol.
* Participants must have been off prior treatment with immunotherapy/investigational agents and chemotherapy for >2 weeks and must have recovered from acute toxicity before the first study treatment administration. Exceptions were participants who needed to receive cytoreductive chemotherapy in order to decrease tumor burden (the study treatment may have started earlier if necessitated by the patient's medical condition (eg, rapidly progressive disease) following discussion with the Sponsor).
* Prior stem cell transplant within 3 months and/or evidence of active systemic Graft versus Host Disease (GVHD) and/or immunosuppressive therapy for GVHD within 1 week before the first study treatment administration.
* Participants with LBL with bone marrow blasts <5%.
* Participants with Burkitt-type ALL.
* Acute leukemia with testicular or central nerve system involvement alone.
* Participants who had developed therapy related acute leukemia.
* Live vaccine(s) within 30 days prior to the first IMP administration or plans to receive such vaccines during the study until 90 days after the last IMP administration.
* Participants with white blood cell count > 50 x10^9/L at the time of screening visit.
* Participants who had been exposed to anti-CD38 therapies within 6 months prior to Day-1.

The above information was not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 28 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2019-08-06 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2023-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (41):
- United States (2):
  - Sarah Cannon Research Institute-Site Number:8400001, Nashville, Tennessee
  - Children's Medical Center of Dallas-Site Number:8400002, Dallas, Texas
- Argentina (4):
  - Investigational Site Number :0320002, CABA, Buenos Aires
  - Investigational Site Number :0320006, Capital Federal, Buenos Aires
  - Investigational Site Number :0320005, Buenos Aires
  - Investigational Site Number :0320004, Buenos Aires
- Brazil (7):
  - Investigational Site Number :0760013, Curitiba, Paraná
  - Investigational Site Number :0760006, Curitiba, Paraná
  - Investigational Site Number :0760007, Porto Alegre, Rio Grande do Sul
  - Investigational Site Number :0760010, Jaú, São Paulo
  - Investigational Site Number :0760009, Ribeirão Preto, São Paulo
  - Investigational Site Number :0760001, São Paulo, São Paulo
  - Investigational Site Number :0760004, São Paulo, São Paulo
- Investigational Site Number :2080001, Copenhagen, Denmark
- France (4):
  - Investigational Site Number :2500002, Lille
  - Investigational Site Number :2500003, Lyon
  - Investigational Site Number :2500001, Paris
  - Investigational Site Number :2500004, Paris
- Germany (3):
  - Investigational Site Number :2760005, Erlangen
  - Investigational Site Number :2760003, Hamburg
  - Investigational Site Number :2760006, Münster
- Investigational Site Number :3000001, Athens, Greece
- Investigational Site Number :3480002, Budapest, Hungary
- Italy (4):
  - Investigational Site Number :3800002, Genoa, Liguria
  - Investigational Site Number :3800001, Monza, Lombardy
  - Investigational Site Number :3800003, Turin, Piedmont
  - Investigational Site Number :3800005, Verona, Veneto
- Mexico (2):
  - Investigational Site Number :4840001, Monterrey, Nuevo León
  - Investigational Site Number :4840005, Col. Rancho Menchaca, Querétaro
- Investigational Site Number :5280001, Utrecht, Netherlands
- Norway (2):
  - Investigational Site Number :5780001, Bergen
  - Investigational Site Number :5780002, Oslo
- Peru (2):
  - Investigational Site Number :6040001, Arequipa
  - Investigational Site Number :6040002, Lima
- Portugal (3):
  - Investigational Site Number :6200002, Coimbra
  - Investigational Site Number :6200001, Lisbon
  - Investigational Site Number :6200003, Porto
- South Korea (3):
  - Investigational Site Number :4100001, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100002, Seoul, Seoul-teukbyeolsi
  - Investigational Site Number :4100004, Seoul, Seoul-teukbyeolsi
- Investigational Site Number :7520001, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- See also: ACT15378 Plain Language Results Summary — https://www.trialsummaries.com/Study/StudyDetails?id=25186&tenant=MT_SNY_9011

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase II, open-label, single-arm study was conducted in 3 separate cohorts at 41 investigational sites in 16 countries. A total of 67 participants were enrolled between 06 Aug 2019 and 08 Jun 2022.
Pre-assignment Details: The study consisted of a screening period (up to 3 weeks prior to the first study treatment administration), treatment period [Day 1 to Day 57 for Acute Lymphoblastic Leukemia(ALL); Day 1 to Day 22 for Acute Myeloid Leukemia(AML)],a period of aplasia followed by recovery period;an end of treatment (EOT) visit within 30 days after hematological recovery and a follow-up period.The study was prematurely stopped due to sponsor decision (stage 2 efficacy criteria not met);not due to safety concerns.
Groups:
- B-cell Acute Lymphoblastic Leukemia (B-ALL): Participants with B-ALL received isatuximab 20 milligram per kilogram (mg/kg) intravenous (IV) infusion once every week (QW) for 4 weeks during the induction period (i.e., on Days 1, 8, 15, and 22) and every 2 weeks (Q2W) during the consolidation period (i.e., on Days 29, 43, and 57. Participants received recommended isatuximab premedication as per protocol. Starting on Day 8, combination chemotherapies were added. Participants without documented disease progression at EOT visit who had not started treatment with another anticancer therapy received follow-up visits every 2 months until initiation of another anticancer therapy, disease progression, death, or final analysis cut-off date, whichever occurred first. Participants with documented disease progression/initiation of new anticancer treatment were followed for survival every 4 months until death or final analysis cut-off date, whichever occurred first.
- T-cell Acute Lymphoblastic Leukemia (T-ALL): Participants with T-ALL received isatuximab 20 mg/kg IV infusion QW for 4 weeks during the induction period (i.e., on Days 1, 8, 15, and 22) and Q2W during the consolidation period (i.e., on Days 29, 43, and 57. Participants received recommended isatuximab premedication as per protocol. Starting on Day 8, combination chemotherapies were added. Participants without documented disease progression at EOT visit who had not started treatment with another anticancer therapy received follow-up visits every 2 months until initiation of another anticancer therapy, disease progression, death, or final analysis cut-off date, whichever occurred first. Participants with documented disease progression/initiation of new anticancer treatment were followed for survival every 4 months until death or final analysis cut-off date, whichever occurred first.
- Acute Myeloid Leukemia (AML): Participants with AML received isatuximab 20 mg/kg IV infusion on Days 1, 8, and 15 of each Cycle (up to 2 treatment cycles, each cycle 28 days). Participants received recommended isatuximab premedication as per protocol. Starting on Day 8, combination chemotherapies were added. Participants without documented disease progression at EOT visit who had not started treatment with another anticancer therapy received follow-up visits every 2 months until initiation of another anticancer therapy, disease progression, death, or final analysis cut-off date, whichever occurred first. Participants with documented disease progression/initiation of new anticancer treatment were followed for survival every 4 months until death or final analysis cut-off date, whichever occurred first.
Period: Overall Study
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Started | 27 | 13 | 27
Completed | 19 | 7 | 20
Not Completed | 8 | 6 | 7
Not completed — Adverse event, not related to Coronavirus Disease-2019 (COVID-19) | 3 | 2 | 3
Not completed — Progressive disease | 5 | 3 | 4
Not completed — Other, Not related to COVID-19 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The All-treated (AT) population consisted of all participants who received at least 1 dose (even incomplete) of study treatment.
Groups:
- B-cell Acute Lymphoblastic Leukemia (B-ALL): Participants with B-ALL received isatuximab 20 mg/kg IV infusion QW for 4 weeks during the induction period (i.e., on Days 1, 8, 15, and 22) and Q2W during the consolidation period (i.e., on Days 29, 43, and 57. Participants received recommended isatuximab premedication as per protocol. Starting on Day 8, combination chemotherapies were added. Participants without documented disease progression at EOT visit who had not started treatment with another anticancer therapy received follow-up visits every 2 months until initiation of another anticancer therapy, disease progression, death, or final analysis cut-off date, whichever occurred first. Participants with documented disease progression/initiation of new anticancer treatment were followed for survival every 4 months until death or final analysis cut-off date, whichever occurred first.
- Total: Total of all reporting groups
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML) | Total
Number analyzed (Participants) | 27 | 13 | 27 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.22 (3.92) | 8.72 (4.15) | 9.04 (5.41) | 8.65 (4.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 4 | 12 | 26
  Male | 17 | 9 | 15 | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 0 | 3
  Asian | 1 | 1 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 2 | 4
  White | 17 | 7 | 15 | 39
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 4 | 4 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response (CR) Rate
Description: The complete response rate (CR + CRi [complete response with incomplete peripheral recovery]) was defined as the percentage of participants achieving complete response (CR + CRi) assessed by the investigator per National Comprehensive Cancer Network (NCCN) guidelines version 1.2018 criteria. CR was defined as <5% blasts in a bone marrow aspirate (BMA) with spicules; no circulating blasts (ALL)/no blasts with Auer rods (AML) or extramedullary disease, no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/central nervous system involvement (ALL), trilineage hematopoiesis (ALL); Absolute neutrophil count (ANC) >=1000/microliter (mcL); platelets >100000/mcL; red blood cell transfusion independence. If the physician documented transfusion dependency related to study treatment and not to the participant's underlying disease, CRi was reported. CRi met the same criteria as for CR, except neutrophils and/or platelets recovery (ANC <1000/mcL or platelets <100000/mcL).
Time Frame: From enrollment until the primary analysis completion date of 12 Sep 2022; the median duration of exposure was approximately 7 weeks
Population: The evaluable population consisted of evaluable participants from the AT population who received at least 1 full dose of isatuximab in Cycle 1 and who had at least 1 valid response value that was evaluable.
Measure: Number; unit: percentage of participants
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
percentage of participants | 52.0 | 45.5 | 60.9

2. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Treatment-Emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant temporally associated with the use of study treatment, whether or not considered related to the study treatment. SAEs were any untoward medical occurrence that at any dose: resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, was a medically important event. TEAEs were defined as an AE which occurred after the first dose of study treatment administration until the last dose plus 30 days, or until the start of hematological recovery period or a new anti-leukemia/lymphoma therapy, whichever occurred first.
Time Frame: From the time of the first treatment administration (Day 1) up to 30 days after the last treatment (maximum duration of exposure of 13.1 weeks for B-ALL cohort, 10.7 weeks for T-ALL cohort and 7.1 weeks for AML cohort)
Population: The AT population consisted of all participants who received at least 1 dose (even incomplete) of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 27 | 13 | 27
Participants
  Any TEAE | 27 | 13 | 26
  Any TESAE | 19 | 12 | 17

3. Secondary Outcome: Number of Participants With Infusion Reactions (IRs)
Description: An IR was an AE related to isatuximab typically with onset within 24 hours from the start of the isatuximab infusion and was reported by the investigator.
Time Frame: as for outcome 2
Population: The AT population consisted of all participants who received at least 1 dose (even incomplete) of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 27 | 13 | 27
Participants | 9 | 5 | 15

4. Secondary Outcome: B-ALL and T-ALL: Area Under the Concentration Time Curve (AUC) of Isatuximab
Description: Plasma samples were collected at specified timepoints to determine the AUC of isatuximab.
Time Frame: From Week 0 to Week 1, Week 0 to Week 5, and Week 0 to Week 10
Population: The Pharmacokinetic (PK) population consisted of all participants from the AT population with at least 1 PK parameter available (isatuximab concentration). Only those participants with data available at specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: mg*hour (h)/Liter (L)
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL)
Number analyzed (Participants) | 27 | 12
mg*hour (h)/Liter (L)
  Week 0 to Week 1 | 31703 (10048) | 29057 (8294)
  Week 0 to Week 5 | 299071 (127581) | 289167 (93095)
  Week 0 to Week 10 | 582686 (316749) | 540375 (233411)

5. Secondary Outcome: AML: AUC of Isatuximab
Description: Plasma samples were collected at specified timepoints to determine the AUC of isatuximab.
Time Frame: From Week 0 to Week 1, Week 0 to Week 3, and Week 0 to Week 8
Population: The PK population consisted of all participants from the AT population with at least 1 PK parameter available (isatuximab concentration). Only those participants with data available at specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: mg*h/L
Arm/Group | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 26
mg*h/L
  Week 0 to Week 1 | 28592 (6858)
  Week 0 to Week 3 | 130862 (40827)
  Week 0 to Week 8 | 291962 (112222)

6. Secondary Outcome: B-ALL and T-ALL: Plasma Concentration Reached by Isatuximab Before Next Dose Administration (Ctrough)
Description: Plasma samples were collected at specified timepoints to determine the Ctrough of isatuximab.
Time Frame: Cycle 1 Day 8, Cycle 1 Day 15, Cycle 1 Day 22, Cycle 1 Day 29, Cycle 2 Day 43, Cycle 2 Day 57
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: microgram/milliliter (mcg/mL)
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL)
Number analyzed (Participants) | 27 | 13
microgram/milliliter (mcg/mL)
  Cycle 1: Day 8: number analyzed (Participants) | 25 | 11
  Cycle 1: Day 8 | 114 (45.7) | 127 (49.9)
  Cycle 1: Day 15: number analyzed (Participants) | 23 | 11
  Cycle 1: Day 15 | 272 (118) | 263 (103)
  Cycle 1: Day 22: number analyzed (Participants) | 15 | 8
  Cycle 1: Day 22 | 388 (163) | 323 (206)
  Cycle 1: Day 29: number analyzed (Participants) | 18 | 9
  Cycle 1: Day 29 | 475 (174) | 426 (209)
  Cycle 2: Day 43: number analyzed (Participants) | 5 | 1
  Cycle 2: Day 43 | 504 (296) | 357 (NA) — Standard deviation (SD) could not be calculated for a single participant.
  Cycle 2: Day 57: number analyzed (Participants) | 8 | 2
  Cycle 2: Day 57 | 531 (224) | 478 (261)

7. Secondary Outcome: AML: Plasma Concentration Reached by Isatuximab Before Next Dose Administration (Ctrough)
Description: Plasma samples were collected at specified timepoints to determine the Ctrough of isatuximab.
Time Frame: Cycle 1 Day 8, Cycle 1 Day 15, Cycle 2 Day 1 and Cycle 2 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 27
mcg/mL
  Cycle 1: Day 8: number analyzed (Participants) | 19
  Cycle 1: Day 8 | 126 (41.0)
  Cycle 1: Day 15: number analyzed (Participants) | 24
  Cycle 1: Day 15 | 217 (60.6)
  Cycle 2: Day 1: number analyzed (Participants) | 10
  Cycle 2: Day 1 | 115 (94.2)
  Cycle 2: Day 15: number analyzed (Participants) | 8
  Cycle 2: Day 15 | 420 (205)

8. Secondary Outcome: B-ALL and T-ALL: Concentrations at the End of Infusion (Ceoi) of Isatuximab
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of isatuximab.
Time Frame: At end of infusion on Cycle 1 Days 1 and 29
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL)
Number analyzed (Participants) | 27 | 13
mcg/mL
  Cycle 1: Day 1: number analyzed (Participants) | 21 | 8
  Cycle 1: Day 1 | 452 (344) | 259 (120)
  Cycle 1: Day 29: number analyzed (Participants) | 19 | 7
  Cycle 1: Day 29 | 835 (366) | 745 (330)

9. Secondary Outcome: AML: Ceoi of Isatuximab
Description: Ceoi is the plasma concentration observed at the end of intravenous infusion of isatuximab.
Time Frame: At end of infusion on Cycle 1 Days 1 and 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 27
mcg/mL
  Cycle 1: Day 1: number analyzed (Participants) | 19
  Cycle 1: Day 1 | 363 (110)
  Cycle 1: Day 15: number analyzed (Participants) | 20
  Cycle 1: Day 15 | 562 (176)

10. Secondary Outcome: Number of Participants With Negative Minimal Residual Disease (MRD)
Description: MRD assessment was performed centrally by next generation sequencing using clonoSEQ and T-cell receptor assays for B-ALL and T-ALL cohorts respectively. It was performed by flow cytometry for AML cohort. Number of participants with CR or CRi who achieved negative MRD in bone marrow and blood was analyzed. In AML indication, peripheral blood tissue is not representative of the tumor burden and cannot be used to assess MRD.
Time Frame: From screening until the study completion date, approximately 45 months
Population: The evaluable population consisted of evaluable participants from the AT population who received at least 1 full dose of isatuximab in Cycle 1 and who had at least 1 valid response value that was evaluable. Only those participants who achieved CR/CRi were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 13 | 5 | 14
Participants
  Blood, 10^-6: number analyzed (Participants) | 13 | 5 | 0
  Blood, 10^-6 | 3 | 1 |
  Bone marrow, 10^-6 | 0 | 2 | 0
  Bone marrow, 10^-3: number analyzed (Participants) | 0 | 0 | 14
  Bone marrow, 10^-3 |  |  | 0

11. Secondary Outcome: Overall Response Rate (ORR)
Description: ORR:Percentage of participants with CR/CRi or partial response (PR) for blood and bone marrow disease based on NCCN guideline. CR: <5% blasts in BMA with spicules; no circulating blasts (ALL)/no blasts with Auer rods (AML) or extramedullary disease, no lymphadenopathy, splenomegaly, skin/gum infiltration/testicular mass/central nervous system involvement (ALL), trilineage hematopoiesis (ALL);ANC >=1000/mcL; platelets >100000/mcL; RBC transfusion independence. If the physician documented transfusion dependency related to study treatment;not to participant's underlying disease, CRi was reported. CRi met the same criteria as CR, except neutrophils and/or platelets recovery (ANC <1000/mcL or platelets <100000/mcL). PR: >50% decrease in the sum of the product of the greatest perpendicular diameters of the mediastinal enlargement. For participants with a previous positive positron emission tomography (PET) scan, a post-treatment PET was to be positive in at least 1 previously involved site.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
percentage of participants | 52.0 [37.5 to 66.2] | 54.5 [31.8 to 75.9] | 65.2 [49.7 to 78.6]

12. Secondary Outcome: Overall Survival (OS)
Description: Overall survival was defined as the time interval from the date of first study treatment administration to death from any cause. It was estimated using the Kaplan-Meier method. Confidence interval (CI) for Kaplan-Meier estimates were calculated with log-log transformation of survival function and methods of Brookmeyer and Crowley.
Time Frame: From first study treatment administration up to death due to any cause, a maximum of 45 months
Population: The evaluable population consisted of evaluable participants from the AT population who received at least 1 full dose of isatuximab in Cycle 1 and who had at least 1 valid response value that was evaluable. Only those participants with data available were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
months | 12.09 [3.975 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 6.85 [2.201 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 9.40 [5.947 to NA] — NA indicates that the upper limit of CI was not estimable due to insufficient number of participants with events at study closure.

13. Secondary Outcome: Event-Free Survival (EFS)
Description: EFS was defined as the time interval from the date of first study treatment administration to the date of the first of: completion or going off protocol induction/consolidation therapy without CR, relapse from CR, or death due to any cause, whichever occurred first. It was estimated using the Kaplan-Meier method. CI for Kaplan-Meier estimates are calculated with log-log transformation of survival function and methods of Brookmeyer and Crowley.
Time Frame: From study treatment administration up to the date of first documented disease progression or death due to any cause, a maximum of 45 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
months | 2.23 [1.413 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 2.14 [1.347 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure. | 5.65 [1.347 to NA] — NA indicates that upper limit of CI was not estimable due to insufficient number of participants with events at study closure.

14. Secondary Outcome: Duration of Response (DoR)
Description: Duration of response was defined as the time from the date of the first response to the date of first disease progression or death from any cause, whichever happens first. It was estimated using the Kaplan-Meier method. CI for Kaplan-Meier estimates are calculated with log-log transformation of survival function and methods of Brookmeyer and Crowley.
Time Frame: From first documented response up to the date of first documented disease progression or death due to any cause, a maximum of 45 months
Population: The evaluable population consisted of evaluable participants from the AT population who received at least 1 full dose of isatuximab in Cycle 1 and who had at least 1 valid response value that was evaluable. Only responders were included in this analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 13 | 5 | 14
months | 7.26 [NA to NA] — Lower and upper limits of CI not estimable due to insufficient number of participants with events at study closure | 1.18 [0.887 to NA] — Upper limit of CI not estimable due to insufficient number of participants with events at study closure | 4.40 [NA to NA] — Lower and upper limits of CI not estimable due to insufficient number of participants with events at study closure

15. Secondary Outcome: Cluster of Differentiation (CD)38 Receptor Density
Description: Blood samples were collected to assess CD38 receptor density as a predictive biomarker. It was assessed across complete responders and non-complete responders. The Antibody Binding Capacity (ABC) was calculated using the following equation: ABC = 10^(Logarithm(Mean Fluorescence Intensity)*a+b) where "a" was the slope and "b" was the Y-intercept of the calibration curve equation. Specific and absolute quantitative values (specific antibody-binding capacity [sABC]) of binding of the selected antibodies were calculated after subtraction of the negative isotypic immunoglobulin G (IgG) control.
Time Frame: Pre-dose on Day 1
Population: The evaluable population consisted of evaluable participants from the AT population who received at least 1 full dose of isatuximab in Cycle 1 and who had at least 1 valid response value that was evaluable. Only those participants with data available at specified timepoints were analyzed.
Measure: Mean (Standard Deviation); unit: sABC
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
sABC
  Blood blast cells: CR/CRi: number analyzed (Participants) | 5 | 2 | 3
  Blood blast cells: CR/CRi | 20345.6 (23439.7) | 12780.0 (15559.2) | 19502.0 (20919.7)
  Blood blast cells: Non CR/CRi;: number analyzed (Participants) | 2 | 1 | 2
  Blood blast cells: Non CR/CRi; | 31080.0 (2397.1) | 22952.0 (NA) — SD cannot be calculated for a single participant. | 9815.0 (4203.0)
  Blood immune cells (Natural Killer [NK] cells): CR/CRi: number analyzed (Participants) | 5 | 2 | 3
  Blood immune cells (Natural Killer [NK] cells): CR/CRi | 13506.2 (3018.6) | 22639.0 (1796.1) | 11220.3 (3764.6)
  Blood immune cells (NK cells): Non CR/CRi: number analyzed (Participants) | 2 | 1 | 2
  Blood immune cells (NK cells): Non CR/CRi | 16650.0 (851.4) | 33859.0 (NA) — SD cannot be calculated for a single participant. | 22530.0 (685.9)

16. Secondary Outcome: CD38 Receptor Occupancy
Description: Blood samples were collected to assess CD38 receptor occupancy as a pharmacodynamics marker. It was assessed across complete responders and non-complete responders. Multicolor flow cytometry assay was validated for CD38 receptor occupancy (CD38RO) quantification, based on the use of two murine monoclonal antibodies (MAbs), one competing with SAR650984 to determine the number of free CD38 receptors (MAb1) and one recognizing a different binding epitope on CD38 to measure the total number of receptors (MAb2) at the cell surface of the cancer cells. Cells were tagged with either MAb1 (Tube #1) or MAb2 (Tube #2). The percentage RO was calculated using the following equation: % CD38RO = [(sABC MAb2 - sABC MAb1)/sABC MAb2] X 100.
Time Frame: Pre-dose on Day 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: percent receptor occupancy
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML)
Number analyzed (Participants) | 25 | 11 | 23
percent receptor occupancy
  Blood plasma cells: CR/CRi: number analyzed (Participants) | 0 | 2 | 0
  Blood plasma cells: CR/CRi |  | 40.5 (30.4) |
  Blood plasma cells: Non CR/CRi;: number analyzed (Participants) | 1 | 1 | 0
  Blood plasma cells: Non CR/CRi; | 44.0 (NA) — SD cannot be calculated for a single participant. | 55.0 (NA) — SD cannot be calculated for a single participant. |
  Blood NK cells: CR/CRi: number analyzed (Participants) | 5 | 3 | 0
  Blood NK cells: CR/CRi | 55.6 (6.9) | 66.7 (2.1) |
  Blood NK cells: Non CR/CRi: number analyzed (Participants) | 3 | 1 | 0
  Blood NK cells: Non CR/CRi | 61.3 (3.5) | 70.0 (NA) — SD cannot be calculated for a single participant. |

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the time of the first treatment administration (Day 1) up to 30 days after the last treatment (maximum duration of exposure of 13.1 weeks for B-ALL cohort, 10.7 weeks for T-ALL cohort and 7.1 weeks for AML cohort). All-cause mortality (Deaths) was collected for the entire study duration, a maximum of 45 months
Description: Analysis was performed on the AT population.
Groups:
- All Participants: All participants in the study were included in this cohort.
Arm/Group | B-cell Acute Lymphoblastic Leukemia (B-ALL) | T-cell Acute Lymphoblastic Leukemia (T-ALL) | Acute Myeloid Leukemia (AML) | All Participants
All-Cause Mortality (participants affected / at risk) | 17/27 | 8/13 | 18/27 | 43/67
Serious Adverse Events (participants affected / at risk) | 19/27 | 12/13 | 17/27 | 48/67
Other Adverse Events (participants affected / at risk) | 26/27 | 12/13 | 24/27 | 62/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-cell Acute Lymphoblastic Leukemia (B-ALL) (N=27) | T-cell Acute Lymphoblastic Leukemia (T-ALL) (N=13) | Acute Myeloid Leukemia (AML) (N=27) | All Participants (N=67)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Bacterial Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Catheter Site Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Disseminated Aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Encephalitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Escherichia Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fournier's Gangrene (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Fungal Infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Fungal Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Genital Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenic Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis Externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumocystis Jirovecii Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Pseudomonal Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 4 (4)
Septic Shock (Infections and infestations) | 3 (3) | 2 (2) | 3 (3) | 8 (8)
Sinusitis Fungal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Staphylococcal Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Febrile Bone Marrow Aplasia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 10 (12) | 5 (6) | 7 (11) | 22 (29)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cytokine Release Syndrome (Immune system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Haemophagocytic Lymphohistiocytosis (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Generalised Tonic-Clonic Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Leukoencephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Cardiac Failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Aortic Aneurysm (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anal Fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Mouth Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Neutropenic Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | B-cell Acute Lymphoblastic Leukemia (B-ALL) (N=27) | T-cell Acute Lymphoblastic Leukemia (T-ALL) (N=13) | Acute Myeloid Leukemia (AML) (N=27) | All Participants (N=67)
Conjunctivitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Device Related Infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Lip Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral Candidiasis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Oral Herpes (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Respiratory Syncytial Virus Infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Skin Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Viral Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (5) | 3 (6)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (6) | 1 (1) | 5 (5) | 10 (12)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Drug Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Food Allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Decreased Appetite (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 8 (8) | 11 (11)
Increased Appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Dysaesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Facial Paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 3 (3) | 3 (4) | 9 (14) | 15 (21)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (2) | 1 (2) | 1 (1) | 4 (5)
Eyelid Oedema (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Periorbital Oedema (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Flushing (Vascular disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 0 (0) | 5 (7) | 3 (3) | 8 (10)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (8) | 1 (1) | 1 (1) | 8 (10)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (5) | 3 (5)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (3)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 2 (2) | 5 (5)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Abdominal Pain (Gastrointestinal disorders) | 6 (6) | 1 (3) | 5 (8) | 12 (17)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Anal Fissure (Gastrointestinal disorders) | 3 (5) | 0 (0) | 2 (2) | 5 (7)
Anal Inflammation (Gastrointestinal disorders) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Colitis (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 5 (5)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (3) | 7 (7) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 3 (3) | 8 (9) | 15 (17)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 4 (6) | 5 (7)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Nausea (Gastrointestinal disorders) | 9 (17) | 3 (5) | 6 (9) | 18 (31)
Oral Pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Stomatitis (Gastrointestinal disorders) | 10 (10) | 4 (5) | 8 (8) | 22 (23)
Vomiting (Gastrointestinal disorders) | 6 (7) | 3 (3) | 10 (15) | 19 (25)
Hepatic Failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic Steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (3) | 3 (4)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 6 (7) | 6 (7)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 2 (6) | 3 (7)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3) | 4 (4)
Bone Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 3 (3)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 4 (6) | 2 (2) | 2 (5) | 8 (13)
Nephropathy Toxic (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Renal Tubular Necrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary Retention (Renal and urinary disorders) | 2 (2) | 3 (4) | 1 (1) | 6 (7)
Catheter Site Pain (General disorders) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Chills (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Face Oedema (General disorders) | 2 (2) | 1 (1) | 0 (0) | 3 (3)
Fatigue (General disorders) | 2 (2) | 1 (1) | 3 (5) | 6 (8)
Oedema Peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 10 (14) | 4 (6) | 12 (23) | 26 (43)
Weight Decreased (Investigations) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Infusion Related Reaction (Injury, poisoning and procedural complications) | 8 (12) | 4 (5) | 14 (16) | 26 (33)

LIMITATIONS AND CAVEATS:
The study was prematurely stopped due to sponsor decision (stage 2 efficacy criteria not met) and not due to safety concerns.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/44/NCT03860844/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT03860844/SAP_001.pdf